CLINICAL TRIAL: NCT04089436
Title: The Threat of Infectious Encephalitis in Southeast Asia: SouthEast Asia Encephalitis Project
Brief Title: SouthEast Asia Encephalitis Project
Acronym: SEAe
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Institut Pasteur (Industry)
Collaborators: Centre De Coopération International En Recherche Agronomique Pour Le Développement (Unknown); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Institut Pasteur, Cambodia (Other); Institut de Recherche pour le Developpement (Other Government); National Institute of Hygiene and Epidemiology, Vietnam (Other); University of Oxford (Other); National Health Laboratory, Myanmar (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2013-024
Record Dates: First submitted 2019-06-28; First posted 2019-09-13 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Encephalitis
Keywords: Encephalitis; Southeast Asia; Japanese encephalitis; Next Generation sequencing
MeSH Terms: conditions — Encephalitis; Encephalitis, Japanese | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — CSF, Whole blood, Buffy Coat, nasopharyngeal and rectal specimen, urine, stool.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with encephalitis: children above 28days and adults with suspected encephalitis Hospitalized in 4 different Hospitals, Kantha Bopha IV children's Hospital, Phnom Penh, Cambodia, National paediatrics Hospital, Hanoi, Vietnam and Mahosot Hospital, Vientiane, Lao PDR, and Yangon Children Hospital, Yangon, Myanmar
  Interventions: Diagnostic Test: CSF sampling; Diagnostic Test: Blood sampling; Diagnostic Test: Nasopharyngeal and rectal sampling

INTERVENTIONS:
Diagnostic Test: CSF sampling — CSF sampling by lumbar puncture
Diagnostic Test: Blood sampling — Blood sampling by blood test
Diagnostic Test: Nasopharyngeal and rectal sampling — Nasopharyngeal and rectal sample by swabbing

SUMMARY:
Encephalitis, an acute inflammation of the central nervous system associated with neurologic dysfunction is of public health concern worldwide, because of its high mortality and neurological sequelae rates. In Asia where many of the possible etiologies are of major public health concerns (i.e. dengue, Japanese encephalitis, West Nile virus, EV71), acute encephalitis is among the most frequent and severe causes of pediatric hospitalization.

Despite extensive microbiological investigations, no pathogen is identified for a significant proportion of encephalitis patients in both industrialized and developing countries (28-85% of cases remain unconfirmed). Unknown and sometimes new emerging infectious agents may be responsible for cases of currently unknown etiology and an intensive effort to identify and characterize them is to be done. From this perspective, the Southeast Asian region, a particularly significant biodiversity hotspot, is at high risk for new pathogen emergence.

Surveillance and diagnostic capabilities for encephalitis remain poor and still suffer from serious shortcomings in most Southeast Asian countries and beyond. Although the burden of non-infectious encephalitis in this region remains to be ascertained, the best laboratories only identify etiological infective agents in less than half of patients. Systematic data regarding the contribution of these diseases are lacking and to define the burden of these infections, to describe the full clinical spectrum and characteristics of acute central nervous system infections, and to develop diagnostic and therapeutic algorithms to improve patient care.

The proposed project is an ambitious and multidisciplinary research consortium that aims to reduce the morbidity and mortality associated with infectious encephalitis in Southeast Asia (Cambodia, Laos, Vietnam and Myanmar) by improving diagnosis and medical care for patients.

The SEAe project specific objectives are:

* To fill-in the biomedical knowledge gaps regarding acute encephalitis syndrome;
* To strengthen hospital laboratories capacities to enhance health by improving diagnosis and care for patients;
* To identify unknown pathogens responsible for encephalitis;
* To provide reliable information and a sustainable regional and sub-regional surveillance network to clinicians and public health stakeholders that will help them to better define prevention policies, vaccination strategy, and build preparedness to emerging infectious risks.

DETAILED DESCRIPTION:
Background:

Encephalitis is defined as an acute inflammation of the central nervous system associated with neurologic dysfunction. The most common etiologies are infections by either viruses or bacteria although parasites and fungi can also be occasionally detected, especially in immunocompromised patients. Because of high mortality and long-term neurological sequelae, encephalitis is of public health concern worldwide. Reported incidences range between 3.5 and 7.4 cases per 100,000 patient-years with higher incidences in children than adults. Various encephalitis outbreaks have recently emerged in Asia such as the fatal outbreak of enterovirus 71 (EV71) that occurred in mid-2012 in Cambodia affecting very young children (most below 3 years, all below 12 years). In Asia where many of the possible etiologies are of major public health concerns (i.e. dengue, Japanese encephalitis, West Nile virus, EV71), acute encephalitis is among the most frequent and severe causes of pediatric hospitalization.

Despite extensive microbiological investigations and the use of the most advanced molecular biology-based assays, no pathogen is identified for a significant proportion of encephalitis patients in both industrialized and developing countries (28-85% of cases remain unconfirmed). Previous studies support the hypothesis that unknown and sometimes new emerging infectious agents may be responsible for cases of currently unknown etiology and strongly argue for an intensive effort to identify and characterize them. This hypothesis is also strengthened by the recent apparent increase in emerging infectious diseases, many of which have been linked to human activities that impact the environment and to the spreading of pathogens to new geographic regions. From this perspective, the Southeast Asian region, a particularly significant biodiversity hotspot, is at high risk for new pathogen emergence. Indeed, growing human populations, increasing urbanization and frequent contact with wildlife and domesticated animals have created novel opportunities for the emergence of pathogens such as SARS at the end of 2002, and highly facilitated the spread of infectious diseases such as H5N1 high-pathogenicity avian influenza virus since 2004, and H1N1 pandemic influenza virus in 2009. The population in developing Southeast Asian countries is particularly at risk for the circulation of emerging or reemerging infectious agents and for this reason the surveillance and investigation of acute encephalitis syndrome in this region is of utmost public health importance, both locally and globally.

Surveillance and diagnostic capabilities for encephalitis remain poor and still suffer from serious shortcomings in most Southeast Asian countries and beyond. Although the burden of non-infectious encephalitis in this region remains to be ascertained, the best laboratories only identify etiological infective agents in less than half of patients. Moreover, because of the absence of reliable microbiological diagnostic capacity in the majority of public referral hospitals, local clinicians have to treat acute encephalitis syndromes mostly empirically, with little evaluation of the effectiveness of their clinical approach. Even if some of the most common causes of acute encephalitis syndrome may be vaccine-preventable, systematic data regarding the contribution of these diseases are lacking and no reliable data are available to define the burden of these infections, to describe the full clinical spectrum and characteristics of acute central nervous system infections, and to develop diagnostic and therapeutic algorithms to improve patient care. Besides, whatever the nature and magnitude of the encephalitis burden in Southeast Asia and the criteria used to assess it (i.e. morbidity, mortality, handicap, impact on families' budget or livelihood), this burden is borne principally by underprivileged populations with limited access to prevention and health care.

Project partners The proposed project is an ambitious and multidisciplinary research consortium associating: (i) national health authorities in Cambodia, Lao PDR, Vietnam and Myanmar; (ii) local major university and clinical sites (national hospitals and provincial health centers); (iii) key French stakeholders of life and health sciences with research activities carried out in the Southeast Asian region such as: Institut Pasteur and the Institut Pasteur International Network, Institut National de la Santé et de la Recherche Médicale (Inserm), Centre de Coopération Internationale en Recherche Agronomique pour le Développement (Cirad), Institut de Recherche pour le Développement (IRD) - Aix-Marseille University - Ecole des Hautes Etudes en Santé Publique (EHESP); and (iv) teams from the Southeast Asian Wellcome Trust Oxford University Major Overseas Programme.

Objectives:

The SEAe project aims to reduce the morbidity and mortality associated with infectious encephalitis in Southeast Asia by improving diagnosis and medical care for patients.

The SEAe project specific objectives are:

* To fill-in the biomedical knowledge gaps regarding acute encephalitis syndrome;
* To strengthen hospital laboratories capacities to enhance health by improving diagnosis and care for patients;
* To identify unknown pathogens responsible for encephalitis;
* To document and analyze factors related to clusters of encephalitis cases integrating human health, animal health and environment through a "One Health" approach;
* To provide reliable information and a sustainable regional and sub-regional surveillance network to clinicians and public health stakeholders that will help them to better define prevention policies, vaccination strategy, and build preparedness to emerging infectious risks.

Population study: patient with suspected encephalitis hospitalized in in 4 different Hospitals, Kantha Bopha IV children's Hospital, Phnom Penh, Cambodia, National paediatrics Hospital, Hanoi, Vietnam and Mahosot Hospital, Vientiane, Lao PDR, Yangon Children Hospital, Yangon, Myanmar. Inclusion criteria were adapted from the International Encephalitis Consortium 2013: all patients should be older than 28 days and presenting an altered mental status (i.e. confusion or inability to talk, decreased or altered level of consciousness or personality change) lasting more than 24 hours without alternative cause identified. These criteria should be associated with at least one of the following: (i) fever (>=38°C axillary) for less than 72 hours before or after presentation; (ii) seizure (febrile seizure excluded); (iii) focal neurologic finding.

Data collection:

Clinical data entries are required for this study.

Data entries:

A single data entry person (a medical doctor) enters clinical information and fill in a paper form at admission, at 24 hours, at discharge and one year after discharge and enter the data into an OpenClinica (hosted in CIRAD server, Montpellier, France ) anonymized online database.

Laboratory data is entered into a customized ACCESS (Microsoft database). The results are entered into dedicated tabs for the different techniques.

A data manager dedicated to the study is in charge of the database. The CIRAD and the Institut Pasteur share the co-ownership of the database.

First statistical analysis will be performed in Institut Pasteur du Cambodge, Phnom Penh, under epidemiology unit responsibility. Continuous data will be described with descriptive statistics, including mean ±SD and/or median (range) as appropriate and categorical data with frequencies (%). Categorical data will be analyzed by univariate analysis with χ2 or Fisher exact test as appropriate and continuous data by nonparametric Mann-Whitney test. Statistical analyses will involve use of R software. Relationships between clinical, biological, radiological variables, etiologies and outcome will be assessed by using a univariate and multivariate logistic regression analyses to identify determinants for poor outcome.

Study Calendar

* Provisional inclusion starting date: July 2014
* Provisional inclusion duration: 3 years and half
* Patient participation duration: 1 year
* Study provisional duration: 5 years
* Data archiving duration: 15 years

ELIGIBILITY:
Inclusion Criteria:

* presenting altered mental status (i.e. confusion or inability to talk, decreased or altered level of consciousness or personality change AND lasting 24 hours or more AND no alternative cause identified);

AND at least one of minor inclusion criteria must be met before patient inclusion:

* presenting fever (38°C axillary) for less than 72 hours before or after presentation;
* seizure (febrile seizure excluded);
* focal neurologic finding.

Exclusion Criteria:

* None

Min Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with suspected encephalitis Hospitalized in 4 different Hospitals, Kantha Bopha IV children's Hospital, Phnom Penh, Cambodia, National paediatrics Hospital, Hanoi, Vietnam and Mahosot Hospital, Vientiane, Lao PDR, and Yangon Children Hospital, Yangon, Myanmar.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2014-07-15 (Actual); Primary Completion 2019-09-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Identify etiologies of encephalitis in South East Asia (Vietnam, Laos, Cambodia and Myanmar). | August 2019
  Proportion of patients with confirmed or probable etiologies and proportion with unidentified pathogen

SECONDARY OUTCOMES:
Describe clinical and biological features of patients with encephalitis | August 2019
  Proportion of participants by demographic data (geographic origin, age), by clinical and biological features assessed by physician (general symptoms, neurological symptoms, length of symptoms, blood pressure, blood pulse, weight, height, white blood cells, platelets counts, hemoglobin, CSF cells, protein glucose levels).
describe clinical outcomes of encephalitis in general and by etiology | December 2019
  Proportion of patient who died or had neurological sequelae or recovered during hospitalization and at one year
Identify factors associated with death or severe neurological sequelea in patients with confirmed infectious encephalitis (survival analyses, sequelea score). | December 2019
  Estimation of risk ratio for death or severe neurological sequelae in patients with confirmed infectious encephalitis by demographic, clinical, and biological data

CONTACTS AND LOCATIONS:
Overall Officials: Marc LECUIT, MD, PhD, Principal Investigator — Institut Pasteur
Locations (7):
- Burma (2):
  - National Health Laboratory, Yangon
  - Yangon children hospital, Yangon
- Cambodia (2):
  - Institut Pasteur of Cambodia, Phnom Penh
  - Kantha Bopha IV children Hospital, Phnom Penh
- Mahidol Oxford Tropical Medicine Research Unit, Vientiane, Laos
- Vietnam (2):
  - National Hospital of Pediatrics, Hanoi
  - National Institute of Hygiene Epidemiology, Hanoi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pommier JD, Gorman C, Crabol Y, Bleakley K, Sothy H, Santy K, Tran HTT, Nguyen LV, Bunnakea E, Hlaing CS, Aye AMM, Cappelle J, Herrant M, Piola P, Rosset B, Chevalier V, Tarantola A, Channa M, Honnorat J, Pinto AL, Rattanavong S, Vongsouvath M, Mayxay M, Phangmanixay S, Phongsavath K, Tin OS, Kyaw LL, Tin HH, Linn K, Tran TMH, Perot P, Thuy NTT, Hien N, Phan PH, Buchy P, Dussart P, Laurent D, Eloit M, Dubot-Peres A, Lortholary O, de Lamballerie X, Newton PN, Lecuit M; SEAe Consortium. Childhood encephalitis in the Greater Mekong region (the SouthEast Asia Encephalitis Project): a multicentre prospective study. Lancet Glob Health. 2022 Jul;10(7):e989-e1002. doi: 10.1016/S2214-109X(22)00174-7. PMID 35714649